CLINICAL TRIAL: NCT01648972
Title: Randomised Double-blind Placebo-controlled Trial of Gastrografin in the Therapeutic Management of Prolonged Postoperative Ileus Following Elective Surgery.
Brief Title: Gastrografin in Postoperative Ileus
Acronym: GAP
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Auckland, New Zealand (Other)
Responsible Party: Principal Investigator, A/Prof Ian Bissett, Associate Professor, University of Auckland, New Zealand
Other Study IDs: UOA-ggRCT1
Record Dates: First submitted 2012-07-24; First posted 2012-07-25 (Estimated); Last update posted 2014-07-04 (Estimated); Status verified 2014-07

CONDITIONS: Prolonged Postoperative Ileus
MeSH Terms: interventions — Diatrizoate Meglumine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gastrografin (Experimental)
  Interventions: Drug: Gastrografin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Gastrografin
  Arms: Gastrografin
Drug: Placebo
  Arms: Placebo

SUMMARY:
After abdominal surgery there is a period of unavoidable dysfunction of the gut. During this time patients are often unable to eat and drink, and do not pass any flatus or stool. Though this resolves within a few days for most, there are a significant number (around 30%) who go on to have a prolonged period of this dysfunction known clinically as postoperative ileus. It has been clearly shown that this group of patients have worse health outcomes and spend a longer time in hospital.

The aim of this study is to trial a drug - gastrografin - in the management of prolonged postoperative ileus. Gastrografin is safe, economical, readily available, and has been used with great success in the similar condition of bowel obstruction. It is predicted that gastrografin will shorten the duration of a prolonged postoperative ileus, thus affording affected patients a better outcome from surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years.
* Current inpatient following elective laparoscopic or open surgery.
* Classified as having prolonged postoperative ileus.
* Able to understand risks/benefits of the study.
* Able to give informed consent.

Exclusion Criteria:

* Pregnancy.
* ASA of 4 or greater.
* Previous allergic reaction to gastrografin or iodinated contrast agents.
* Manifest hyperthyroidism.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2012-09; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Time from diagnosis (and administration of study drug) to resolution of prolonged postoperative ileus.

SECONDARY OUTCOMES:
Length of hospital stay (days) | Days

CONTACTS AND LOCATIONS:
Locations (1):
- Auckland City Hospital, Auckland, AKL, New Zealand